CLINICAL TRIAL: NCT01446406
Title: Electronic Daily Self-monitoring of Subjective and Objective Symptoms in Bipolar Disorder - The MONARCA Project (MONitoring, treAtment and pRediCtion of bipolAr Disorder Episodes)
Brief Title: The MONARCA Project (MONitoring, treAtment and pRediCtion of bipolAr Disorder Episodes)
Acronym: MONARCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Centre Rigshospitalet (Other)
Collaborators: University of Copenhagen (Other); IT University of Copenhagen (Other); The European Union, 7.th Frame program (Unknown)
Responsible Party: Principal Investigator, Maria Faurholt-Jepsen, Principal Investigator, Medical doctor and PhD student, Psychiatric Centre Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2011-056
Record Dates: First submitted 2011-09-26; First posted 2011-10-05 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Electronic daily monitoring; Affective episodes
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MONARCA (Active Comparator): MONARCA self-monitoring application on a cell phone to monitor affective symptoms every day.
  Interventions: Device: MONARCA
- NON-MONARCA (Placebo Comparator): This is the same mobile phone as the MONARCA mobile phone. Yet the MONARCA application has not been installed. The mobile phone can only be used as a normal mobile phone for communication purposes.
  Interventions: Device: NON-MONARCA

INTERVENTIONS:
Device: MONARCA — Monitoring affective symptoms entered by the patient every day.
  Other Names: Electronic self-monitoring
  Arms: MONARCA
Device: NON-MONARCA — A mobile phone for communication purposes only. No application has been installed.
  Arms: NON-MONARCA

SUMMARY:
Bipolar disorder is associated with a high risk of relapse and hospitalisation and many patients do not recover to previous psychosocial function. Major reasons for poor outcome are delayed intervention for prodromal depressive and manic episodes as well as decreased adherence with treatment. Recently, electronic self monitoring of affective symptoms using cell phones to prompt patients to respond to weekly text messages has been suggested as an easy and cheap way to identify early signs of affective episodes. Nevertheless, so far the electronic devises has been rather simple not including a bi-directional feed back loop between patients and providers and without electronic data on "objective" measures of the affective psychopathology. As part of an ongoing EU research program a software program for online electronic self-monitoring using a cell phone is being developed including an interactive feed back loop between patients, relatives and clinicians. Electronic self-monitoring includes subjective items such as mood, irritability, sleep duration, activity, alcohol consumption, medication intake and objective items of speech duration (on the cell phone), social activity (numbers of calls and SMS'es at the cell phone) and physical activity (acceleration of the cell phone). The present PhD. study will in a randomized controlled single blind trial including 60 patients with bipolar disorder allocated to using the active cell phone program (intervention group) or to using a cell phone to usual communication (control group) during a 6 months study period.

If the cell phone self-monitoring system is proved effective in preventing mood symptoms and improving psychosocial functioning,quality of life etc. in the present study there might be basis for extending the use of the system to treatment of patients with bipolar disorder in clinical practice in general.

DETAILED DESCRIPTION:
The objectives of the study are to investigate in a randomised controlled single blind trial whether the use of an online monitoring system in patients suffering from bipolar disorder reduces symptoms of affective disorder.

As part of the clinical assessment in the Mood Disorder clinic, a paper version with daily monitoring of subjective items has been in use for four years. Based on an interactive process with patients suffering from bipolar disorder, the literature as well as clinical experience of the research and clinical group involved in the study we have chosen to monitor the following subjective items: mood, activity, irritability, sleep duration, alcohol consumption, medication intake. Patients are prompted to evaluate these items every evening. In the same way, the following objective items will be collected on all cell phones used in the study: speech duration (minutes speech per 24 hours on the cell phone), social activity (numbers of calls and SMS'es per 24 hours at the cell phone and acceleration of the cell phone).

A personal homepage for each patient is set op on a server so the patient can connect to the homepage with his cell phone using secure codes. By giving informed consent to participate in the MONARCA trial patients allow clinicians to connect to the homepage. It is optionally whether patients allow relatives (or others) to get access to the homepage. Online programs present the monitored subjective items as well as speech duration and number of calls and SMS's graphically.

It is not known whether using a cell phone for electronic monitoring of bipolar disorder the way described above improve outcome compared to using a cell phone to usual communication. A total of 60 patients with bipolar disorder are randomised (1:1) to using the active cell phone program (intervention group) or to using a cell phone to usual communication (control group). All randomised patients will receive a cell phone (Android) for use during the study period.

Stratification is done for age (18-30 versus 30-60 years) and prior hospitalisations (none versus hospitalisation). Study period: 6 months

The assessments are done by the PhD.-student who is not involved in the treatment of the randomised patients and is blinded versus having received the intervention system or the control system. All participants in the study will be examined every month by the PhD student for the entire study period. The following will be done: The bipolar diagnosis is confirmed by a SCAN interview. Further the following ratings/questionnaires are performed every month for 6 months: Hamilton Depression Scale-17 items (HAMD-17), the Young Mania Rating Scale (YMRS), psychosocial functioning (FAST), Cohen's Perceived stress scale, quality of life (WHOQOL), coping strategies (CISS), Altman Self-rating mania scale, Major Depression Inventory (MDI). Assessment of cognitive function (SCIP and Massachusetts General Hospital Questionnaire), awakening salivary cortisol, urinary oxidative stress, adherence to medication (plasma values of medication) and plasma BDNF are measured at start, half way and end of the study.

All assessment is done single blind, i.e., the assessor (researcher) does not know whether the patient is randomized to the intervention group or the control group.

The outcomes are differences between intervention and control group in:

* Primary: depressive and manic symptoms
* Secondary: psychosocial functioning, quality of life, perceived stress, coping strategies,adherence to medication, cognitive function, awakening salivary cortisol, urinary oxidative stress, plasma BDNF, physical activity, self-rated depressive and manic symptoms

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar disorder
* Hamilton Depression Scale under or equal to 17
* Young Mania Rating Scale under or equal to 17

Exclusion Criteria:

* Significant somatic disease
* Other severe mental illness (schizophrenia, schizoaffective disorder)
* Lack of technical skills
* Lack of knowledge of Danish
* Pregnancy
* Lack of desire/willingness to use the delivered cell phone as primary phone

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2011-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Differences in Hamilton Depression Rating Scale (HAM-D17) score and Young Mania Rating Scale (YMRS) score during the entire 6 months study period. | Measured on all participants included one time a month for six months
  The differences in scores on HAM-D17 and YMRS in the areas under the curves between the intervention and the control group.

SECONDARY OUTCOMES:
Psychosocial Functioning (Functioning Assessment Short Test, FAST) | Measured every month for 6 months on all participants
  Differences between the two groups in: psychosocial functioning, quality of life, perceived stress, coping strategies,adherence to medication, cognitive function, awakening salivary cortisol, urinary oxidative stress, plasma BDNF, physical activity, self-rated depressive and manic symptoms (secondary)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Faurholt-Jepsen, MD, Principal Investigator — Department of psychiatry, Copenhagen, Denmark
Locations (1):
- Psychiatric Center Copenhagen, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Faurholt-Jepsen M, Frost M, Christensen EM, Bardram JE, Vinberg M, Kessing LV. Validity and characteristics of patient-evaluated adherence to medication via smartphones in patients with bipolar disorder: exploratory reanalyses on pooled data from the MONARCA I and II trials. Evid Based Ment Health. 2020 Feb;23(1):2-7. doi: 10.1136/ebmental-2019-300106. PMID 32046986
- [Derived] Faurholt-Jepsen M, Vinberg M, Christensen EM, Frost M, Bardram J, Kessing LV. Daily electronic self-monitoring of subjective and objective symptoms in bipolar disorder--the MONARCA trial protocol (MONitoring, treAtment and pRediCtion of bipolAr disorder episodes): a randomised controlled single-blind trial. BMJ Open. 2013 Jul 24;3(7):e003353. doi: 10.1136/bmjopen-2013-003353. Print 2013. PMID 23883891